CLINICAL TRIAL: NCT00409942
Title: Prospective, Randomised, Open, Blinded-endpoint Study of Torasemide Prolonged Release vs Furosemide to Evaluate the Efficacy on Myocardial Fibrosis in Patients With Heart Failure
Brief Title: Effect of a New Formulation of Torasemide (Prolonged Release)on Myocardial Fibrosis in Patients With Heart Failure.
Acronym: TORAFIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Savion Gropper, ferrer
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N/GF-TORAFIC-06; EudraCT number 2006-001446-14
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-06

CONDITIONS: Congestive Heart Failure
Keywords: Chronic heart failure; Torasemide prolonged release; Myocardial fibrosis; Loop diuretics; Peptide of procollagen type 1
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Torasemide prolonged released
  Interventions: Drug: Torasemide Prolonged Release
- 2 (Active Comparator): Furosemide
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Torasemide Prolonged Release — Torasemide Prolonged release 10mg/day up to 40mg/day, treatment duration:8 months
  Other Names: Torasemide Prolonged release:Sutril neo
  Arms: 1
Drug: Furosemide — Furosemide 40mg/day up to 160mg/day, Treatment duration:8 months
  Other Names: Furosemide: Seguril
  Arms: 2

SUMMARY:
Torasemide is a loop diuretic (pyridine-sulfonylurea)with a wide experience in the treatment of oedema associated to heart failure, kidney or liver disease and either in the treatment of arterial hypertension (alone or combined with other anti-hypertensive drugs). It has been developed a new formulation of Torasemide (Torasemide prolonged release).

The aim of this trial is to study the effects of Torasemide prolonged released in comparison with furosemide, in the reduction of myocardial fibrosis in patients with chronic heart failure (Class II-IV of the New York Heart Association Classification.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Patients with chronic heart failure class II-IV (NYHA)due to arterial hypertension
* Patients clinically stable who required diuretic treatment
* Patients with left ventricular hypertrophy diagnosed by echocardiogram
* Patients without ischaemic cardiopathy or non recent disease
* Signed Informed Consent

Exclusion Criteria:

* Heart Failure due to aortic stenosis or hypertrophic myocardiopathy
* Recent coronary syndrome (less than 3 months)
* Recent myocardial infarction (less than 6 months)
* Unstable angor pectoris
* Severe cardiac arrhythmia
* Pregnancy or breastfeeding
* Aldosterone antagonists (last 6 months)
* Current loop diuretic treatment over study doses (torasemide > 10mg/day furosemide > 40 mg/day)
* known hypersensitivity to study drugs
* Liver disease (SGPT or AST > twice upper normal limt)
* Renal impairment (Serum creatinine > 2,5mg/dl)
* Insulin-dependent diabetes
* Patient included in another simultaneous study
* Lactose intolerance
* Lithium Concomitant treatment
* Chronic treatment with NSAIDs
* Concomitant treatment with aminoglycoside antibiotics,etacrynic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Myocardial fibrosis reduction:measure of Serum carboxy-terminal peptide of procollagen type 1. | 8 months

SECONDARY OUTCOMES:
Clinical improvement (New York Heart Association classification, signs and symptoms of heart failure) | 8 months
Cardiovascular events | 8 months
NT-proBNP (Brain Natriuretic Peptide) | 8 months
Hospitalizations, home care due to cardiovascular causes related to heart failure | 8 months
Safety and tolerability | 8 months
Quality of Life (Minnesota Test) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Coca, MD, PhD, Study Chair — Hospital Clinic of Barcelona; Manuel Anguita, MD, PhD, Study Chair — Hospital Reina Sofia - Córdoba; Eduardo De Teresa, MD, PhD, Study Chair — Hospital Clinico - Málaga; Alfonso Castro Beiras, MD, PhD, Study Chair — Hospital Juan Canalejo - Coruña; Javier Díez, Study Director — Centro Investigación Médica Aplicada (CIMA) - Pamplona (Navarra)
Locations (23):
- Spain (23):
  - Clinc Hospital, Barcelona, Barcelona
  - Germans Trias i Pujol Hospital, Barcelona, Barcelona
  - H. del Mar, Barcelona, Barcelona
  - Valle Hebrón Hospital, Barcelona, Barcelona
  - Canet de Mar, Primary Care Centre, Canet de Mar, Barcelona
  - Centelles - Primar Care Centre, Centellas, Barcelona
  - El Maresme - Primary Care Centre, Mataró, Barcelona
  - Remei, Primary care centre, Vic, Barcelona
  - Reina Sofia Hospital, Córdoba, Córdoba
  - Josep Trueta Hospital, Girona, Girona
  - San Jorge Hospital, Huesca, Huesca
  - Complejo Hospitalario Juan Canalejo, A Coruña, La Coruña
  - Begonte - Primary Care Centre, Begonte, Lugo
  - Gregorio Marañón Hospital, Madrid, Madrid
  - Clinico Universitario Virgen de la Victoria, Málaga, Malaga
  - Virgen de la Arrixaca, Murcia, Murcia
  - Central Hospital, Oviedo, Principality of Asturias
  - Clinico Universitario Hospital, Salamanca, Salamanca
  - Donostia Hospital, Donostia / San Sebastian, San Sebastián
  - Clinico Universitario de Santiago, Santiago de Compostela, Santiago de Compostela
  - Alcover - primary care centre, Alcover, Tarragona
  - General Hospital, Valencia, Valencia
  - Clinico Universitario, Zaragoza, Zaragoza

REFERENCES:
- [Background] Querejeta R, Lopez B, Gonzalez A, Sanchez E, Larman M, Martinez Ubago JL, Diez J. Increased collagen type I synthesis in patients with heart failure of hypertensive origin: relation to myocardial fibrosis. Circulation. 2004 Sep 7;110(10):1263-8. doi: 10.1161/01.CIR.0000140973.60992.9A. Epub 2004 Aug 16. PMID 15313958
- [Background] Gonzalez A, Lopez B, Diez J. New directions in the assessment and treatment of hypertensive heart disease. Curr Opin Nephrol Hypertens. 2005 Sep;14(5):428-34. doi: 10.1097/01.mnh.0000174143.30045.bd. PMID 16046900
- [Background] Lopez B, Querejeta R, Gonzalez A, Sanchez E, Larman M, Diez J. Effects of loop diuretics on myocardial fibrosis and collagen type I turnover in chronic heart failure. J Am Coll Cardiol. 2004 Jun 2;43(11):2028-35. doi: 10.1016/j.jacc.2003.12.052. PMID 15172408
- [Background] Lopez B, Gonzalez A, Querejeta R, Diez J. The use of collagen-derived serum peptides for the clinical assessment of hypertensive heart disease. J Hypertens. 2005 Aug;23(8):1445-51. doi: 10.1097/01.hjh.0000173780.67308.f1. PMID 16003166
- [Background] Lopez B, Gonzalez A, Beaumont J, Querejeta R, Larman M, Diez J. Identification of a potential cardiac antifibrotic mechanism of torasemide in patients with chronic heart failure. J Am Coll Cardiol. 2007 Aug 28;50(9):859-67. doi: 10.1016/j.jacc.2007.04.080. Epub 2007 Aug 13. PMID 17719472
- [Derived] TORAFIC Investigators Group. Effects of prolonged-release torasemide versus furosemide on myocardial fibrosis in hypertensive patients with chronic heart failure: a randomized, blinded-end point, active-controlled study. Clin Ther. 2011 Sep;33(9):1204-1213.e3. doi: 10.1016/j.clinthera.2011.08.006. Epub 2011 Sep 8. PMID 21906812
- [Derived] Diez J, Coca A, de Teresa E, Anguita M, Castro-Beiras A, Conthe P, Cobo E, Fernandez E; TORAFIC Investigators Group. TORAFIC study protocol: torasemide prolonged release versus furosemide in patients with chronic heart failure. Expert Rev Cardiovasc Ther. 2009 Aug;7(8):897-904. doi: 10.1586/erc.09.74. PMID 19673667